CLINICAL TRIAL: NCT01646255
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of The Efficacy And Safety of Rotigotine Transdermal Patch In Chinese Subjects With Advanced-stage, Idiopathic Parkinson's Disease Who Are Not Well Controlled On Levodopa
Brief Title: Rotigotine Versus Placebo, A Study To Evaluate The Efficacy In Advanced Stage Idiopathic Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: UCB Trading (Shanghai) Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP1037
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Rotigotine; Neupro phase 3; Advanced-stage; Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine; Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine, daily doses, treatment group
  Interventions: Drug: Rotigotine; Drug: L-dopa
- Placebo (Placebo Comparator): Placebo, daily doses, placebo group
  Interventions: Drug: Placebo Patch; Drug: L-dopa

INTERVENTIONS:
Drug: Rotigotine — Transdermal Patch
  Content:
  4 mg /24 h (20 cm^2), 6 mg /24 h (30 cm^2), 8 mg /24 h (40 cm^2)
  For advanced-stage Parkinson's Disease, subjects received Rotigotine patches in escalating weekly dose (starting with daily doses 4 mg/24 h to 16 mg/24 h) for a maximum 7-week Titration Period, then 12 week maintenance period
  Arms: Rotigotine
Drug: Placebo Patch — Transdermal Patch
  Size:
  20 cm^2, 30 cm^2, 40 cm^2
  Subjects randomized to placebo received matching placebo patches
  Arms: Placebo
Drug: L-dopa — Subject must be on a stable dose of L-dopa (either short-acting or sustained release [in combination with benserazide or carbidopa]) of at least 200 mg/day, administered in at least 2 intakes, for at least 28 days prior to Baseline.
  Other Names: Levodopa

SUMMARY:
The primary objective of this study was to demonstrate that Rotigotine transdermal patch is efficacious in Chinese subjects with advanced-stage Idiopathic Parkinson's Disease as an adjuvant therapy.

DETAILED DESCRIPTION:
The study included a maximum 4-week Screening Period, a maximum 7-week Titration Period for advanced-stage Parkinson's disease, 12-week Maintenance Period, a maximum 12-day De-escalation Period for advanced-stage Parkinson's Disease and 30-day Safety Follow-Up Period. The maximum study duration for an individual subject with advanced-stage Parkinson's disease was 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* An Independent Ethics Committee (IEC)-approved written informed consent is signed and dated by the subject or by the legal representative
* Subject/legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and medication application according to the judgment of the investigator
* Subject has Idiopathic Parkinson's Disease of more than 3 years' duration, defined by the cardinal sign, Bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes, and without any other known or suspected cause of Parkinsonism
* The investigator must observe the subject in both the 'on' and 'off' state and determine that the subject is Hoehn & Yahr stage 2 through 4 in both the 'on' and 'off' state
* Subject is male or female and aged ≥30 years at Screening (Visit 1)
* Subject has a Mini Mental State Examination (MMSE) score of ≥25 at Screening (Visit 1)
* Subject must be on a stable dose of L-dopa (either short-acting or sustained release [in combination with Benserazide or Carbidopa]) of at least 200 mg/day, administered in at least 2 intakes, for at least 28 days prior to Baseline (Visit 2)
* Subject is not adequately controlled on a L-dopa dose (in combination with Benserazide or Carbidopa) which was judged by the treating physician to be optimal
* Subject must be willing and able to accurately complete a subject diary on designated days (with assistance from caregivers, if required), recording periods when they are 'on without troublesome Dyskinesia', 'on with troublesome Dyskinesia', 'off', and sleeping
* As part of the Screening (pretreatment) assessments, the subject must complete a diary over a period of 6 days, with 4 of the 6 diaries being 'valid' as determined by the investigator (see Section 9.1.1)
* It must be clear to the investigator that the subject is able to differentiate between the 'on' and 'off' state and the 'valid' diaries confirm that the subject has an average of ≥2.5 h/day spent in the 'off' state
* If the subject is receiving an Anticholinergic agent (eg, Benztropine, Trihexyphenidyl, Parsitan, Procyclidine, Biperiden), a monoamine oxidase (MAO)-B inhibitor (eg, Selegiline), and/or an N-methyl-d-aspartate (NMDA) antagonist (eg, Amantadine), he/she must have been on a stable dose for at least 28 days prior to Baseline (Visit 2) and be maintained on that dose for the duration of the study
* Subject must be on a stable dose of all anti-Parkinsonian medications for at least 20 days prior to completing the 6 Baseline diaries

Exclusion Criteria:

* Subject has previously participated in this study or subject has previously received the study medication under investigation in this study
* Subject is participating in another study of an investigational drug or has done so within 28 days prior to the Baseline Visit (Visit 2)
* Subject has a history of significant skin hypersensitivity to adhesive or other transdermal preparations, or recent unresolved contact dermatitis
* Subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1)
* Subject has atypical Parkinson's syndrome(s) due to drugs (eg, Metoclopramide, Flunarizine), Metabolic Neurogenetic Disorders (eg, Wilson's Disease), Encephalitis, Cerebrovascular Disease, or Degenerative Disease (eg, Progressive Supranuclear Palsy)
* Subject has a history of Pallidotomy, Thalamotomy, deep brain stimulation, or fetal tissue transplant
* Subject has dementia, active psychosis or hallucinations, or severe depression
* Subject is receiving therapy with a Dopamine agonist either concurrently or has done so within 28 days prior to the Baseline Visit (Visit 2)
* Subject is receiving therapy with 1 of the following drugs either concurrently or within 28 days prior to Baseline (Visit 2): Alpha-methyl dopa, Metoclopramide, Reserpine, Neuroleptics (except specific atypical neuroleptics: Olanzapine, Ziprasidone, Aripiprazole, Clozapine, quetiapine), MAO-A inhibitors, Methylphenidate, or Amphetamine
* Subject is currently receiving central nervous system (CNS) active therapy (eg, sedatives, hypnotics, antidepressants, anxiolytics), unless the dose has been stable for at least 28 days prior to Baseline (Visit 2) and is likely to remain stable for the duration of the study
* Subject has a current diagnosis of Epilepsy, has a history of seizures as an adult, has a history of stroke, or has had a transient ischemic attack within 1 year prior to Screening (Visit 1)
* Subject has clinically relevant hepatic dysfunction (as defined as a total bilirubin >2.0 mg/dL, or Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) >2 times the upper limit of the reference range)
* Subject has clinically relevant renal dysfunction (serum creatinine >2.0 mg/dL [>178 μmol/L])
* Subject has clinically relevant cardiac dysfunction (any cardiac disorder which in the opinion of the investigator would put the subject at risk of clinically relevant arrhythmia) and/or myocardial infarction within the last 12 months
* Subject has a QT interval corrected for heart rate according to Bazett's formula (QTcB) of ≥500 ms at Screening (Visit 1)
* Subject has a history of only symptomatic (not asymptomatic) orthostatic hypotension, with a decrease of systolic blood pressure (SBP) from supine to standing position of ≥2 0 mmHg or of ≥10 mmHg in DBP after 1 or 3 minutes within 28 days prior to Baseline (Visit 2), or SBP <105 mmHg at study entry 17. Subject has evidence of an impulse control disorder (ICD) at Screening (Visit 1)
* Subject has a history of known intolerance/hypersensitivity to the following Antiemetics: Domperidone, Trimethobenzamide, Ondansetron, Tropisetron, Granisetron, and Glycopyrrolate
* Subject has a history of chronic alcohol or drug abuse within the last 5 years
* Subject is pregnant or nursing, or is of childbearing potential but (i) not surgically sterile or (ii) not using adequate birth control methods (including at least a double barrier method) or (iii) not sexually abstinent or (iv) not at least 2 years post-menopausal
* Subject has any other clinically relevant medical condition, psychiatric condition, or laboratory abnormality which would, in the judgment of the investigator, interfere with the subject's ability to participate in the study

Exclusion Criteria:

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1 877 822 9493
Locations (24):
- China (24):
  - Sp1037 001, Beijing
  - Sp1037 002, Beijing
  - Sp1037 019, Beijing
  - Sp1037 025, Beijing
  - Sp1037 017, Changchun
  - Sp1037 007, Chengdu
  - Sp1037 027, Chengdu
  - Sp1037 021, Fuzhou
  - Sp1037 010, Guangzhou
  - Sp1037 011, Guangzhou
  - Sp1037 014, Guangzhou
  - Sp1037 015, Guangzhou
  - Sp1037 005, Hangzhou
  - Sp1037 013, Hangzhou
  - Sp1037 018, Hangzhou
  - Sp1037 023, Jinan
  - Sp1037 003, Shanghai
  - Sp1037 004, Shanghai
  - Sp1037 009, Shanghai
  - Sp1037 008, Suzhou
  - Sp1037 016, Tianjin
  - Sp1037 006, Wuhan
  - Sp1037 022, Wuhan
  - Sp1037 024, Wuhan

REFERENCES:
- [Result] Zhang ZX, Liu CF, Tao EX, Shao M, Liu YM, Wang J, Asgharnejad M, Xue HB, Surmann E, Bauer L. Rotigotine transdermal patch in Chinese patients with advanced Parkinson's disease: A randomized, double-blind, placebo-controlled pivotal study. Parkinsonism Relat Disord. 2017 Nov;44:6-12. doi: 10.1016/j.parkreldis.2017.08.015. Epub 2017 Aug 10. PMID 28827011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, randomized, double-blind, parallel-group, placebo-controlled study started recruiting in August 2012.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS), consisting of all randomized subjects who received at least 1 dose of study medication.
Groups:
- Placebo: Subjects randomized to placebo received matching placebo patches.
- Rotigotine: Subjects received rotigotine in escalating weekly doses (starting with daily doses of rotigotine 4 mg/ 24 h or matching placebo) until an optimal dose or maximal dose of rotigotine 16 mg/ 24 h was achieved. Each dose level was maintained for 1 week.
Period: Overall Study
Arm/Group | Placebo | Rotigotine
Started | 172 | 174
Completed | 151 | 160
Not Completed | 21 | 14
Not completed — Adverse Event | 7 | 8
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 10 | 6
Not completed — Compliance is not well | 1 | 0
Not completed — Inclusion Criteria Deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refers to to the Safety Set (SS), consisting of all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Placebo | Rotigotine | Total Title
Number analyzed (Participants) | 172 | 174 | 346
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 96 | 111 | 207
  >=65 years | 76 | 63 | 139
Age, Continuous [Mean (Standard Deviation); unit: years]
  mean (standard deviation) | 62.8 (9.1) | 61.7 (8.8) | 62.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 81 | 143
  Male | 110 | 93 | 203
Weight [Mean (Standard Deviation); unit: kg] | 61.83 (10.18) | 60.38 (10.15) | 61.10 (10.18)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Absolute Time Spent 'Off' From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "off" when he/she began to lose the optimum effects of anti-Parkinson's medication. A negative mean indicates a reduction of the time off during the conduct of the study
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: The Full Analysis Set (FAS) consisted of all subjects who have been randomized, received at least 1 dose of study medication, had a valid Baseline primary efficacy measurement, and had at least 1 valid post-Baseline primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Full Analysis Set (Placebo Treated Subjects): Subjects randomized to placebo received matching placebo patches.
- Full Analysis Set (Rotigotine Treated Subjects): Subjects received rotigotine in escalating weekly doses (starting with daily doses of rotigotine 4 mg/ 24 h or matching placebo) until an optimal dose or maximal dose of rotigotine 16 mg/ 24 h was achieved. Each dose level was maintained for 1 week.
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
hours | -1.13 (3.20) | -2.36 (2.83)
Statistical Analysis 1: Comparison: Full Analysis Set (Placebo Treated Subjects) vs Full Analysis Set (Rotigotine Treated Subjects); Estimate of treatment effect has been obtained from an analysis of covariance (ANCOVA) model to the change from Baseline value in absolute time spent "off". The ANCOVA model contained treatment and (pooled) site as factors and Baseline "off" time as covariate. A last observation carried forward (LOCF) imputation approach was used for missing values (during both Titration and Maintenance Periods) for the primary efficacy analysis; Test type: Superiority or Other; p = 0.0002, ANCOVA — Primary efficacy analyses was made with confirmatory 2-sided test with significance level 0.05; Least Square Mean = -1.20, 95% CI 2-sided [-1.83 to -0.57]

2. Secondary Outcome: Percentage of Responders From Baseline to the End of the Doubleblind Maintenance Period
Description: A Responder is defined as a subject with an ≥ 30 % decrease in absolute time spent 'off'
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Full Analysis Set (Rotigotine Treated Subjects): Subjects received rotigotine patches in escalating weekly doses (starting with daily doses of rotigotine 4 mg/ 24 h) until an optimal dose or maximal dose of rotigotine 16 mg/ 24 h or matching placebo was achieved. Each dose level was maintained for 1 week.
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percentage of participants | 36.9 | 48.8

3. Secondary Outcome: Percent Change in Absolute Time Spent "Off" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "off" when he/she began to lose the optimum effects of anti-Parkinson's medication.
  Absolute time "off" is defined as the mean number of hours marked "off" during a 24-hour period from all valid daily diary cards.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percent change | -15.0 (56.56) | -36.03 (43.03)

4. Secondary Outcome: Percent Change in Relative Time Spent "Off" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "off" when he/she began to lose the optimum effects of anti-Parkinson's medication.
  Relative time spent "off" will be calculated in two stages. Each valid daily diary will have an associated relative time "off" calculated as relative time "off" for day = 100*[total absolute time "off" for day/ absolute time awake for day]. Relative time spent "off" is then calculated by averaging the daily relative time "off" for the valid days of that visit.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percent change | -14.86 (53.26) | -34.97 (43.87)

5. Secondary Outcome: Change in Absolute Time Spent "on" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was 'off' when taking his/her L-dopa, he/she recorded the exact time their status changed to 'on'.
  Absolute time "on" is defined as the mean number of hours marked "on" during a 24-hour period from all valid daily diary cards.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
hours | 0.94 (3.08) | 2.05 (2.98)

6. Secondary Outcome: Change in Relative Time Spent "on" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was "off" when taking his/her L-dopa, he/she recorded the exact time their status changed to "on".
  Relative time spent "on" will be calculated in two stages. Each valid daily diary will have an associated relative time "on" calculated as relative time "on" for day = 100*[total absolute time "on" for day/ absolute time awake for day]. Relative time spent "on" is then calculated by averaging the daily relative time "on" for the valid days of that visit.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
hours | 6.78 (19.61) | 14.49 (18.70)

7. Secondary Outcome: Percent Change in Absolute Time Spent "on" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was 'off' when taking his/her L-dopa, he/she recorded the exact time their status changed to 'on'.
  Note for percent change calculations: when absolute time at Baseline was 0 hours, the absolute Baseline value was assumed to be 1 minute for calculation purposes.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percent change | 13.53 (42.74) | 368.55 (4446.55)

8. Secondary Outcome: Percent Change in Relative Time Spent "on" From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was "off" when taking his/her L-dopa, he/she recorded the exact time their status changed to "on".
  Note for percent change calculations: when relative time at Baseline was 0%, the relative Baseline value was assumed to be 0.1 for calculation purposes.
  Relative time spent "on" will be calculated in two stages. Each valid daily diary will have an associated relative time "on" calculated as relative time "on" for day = 100*[total absolute time "on" for day/ absolute time awake for day]. Relative time spent "on" is then calculated by averaging the daily relative time "on" for the valid days of that visit.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percent change | 14.99 (42.60) | 616.80 (7667.58)

9. Secondary Outcome: Change in the Number of "Off" Periods From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "off" when he/she began to lose the optimum effects of anti-Parkinson's medication.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of 'off' Periods
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
Number of 'off' Periods | -0.61 (1.59) | -0.89 (1.32)

10. Secondary Outcome: Change in Status of the Subject (on) After Wake-up With Troublesome Dyskinesia From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was 'off' when taking his/her L-dopa, he/she recorded the exact time their status changed to 'on'.
  The percentage of days from Baseline to the end of the double-blind Maintenance Period in which the subject woke in the "on with troublesome dyskinesia" state is presented below.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percentage of days | 2.42 (21.70) | 1.24 (16.90)

11. Secondary Outcome: Change in Status of the Subject (on) After Wake-up Without Troublesome Dyskinesia From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was 'off' when taking his/her L-dopa, he/she recorded the exact time their status changed to 'on'.
  The percentage of days from Baseline to the end of the double-blind Maintenance Period in which the subject woke in the "on without troublesome dyskinesia" state is presented below.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percentage of days | 7.92 (43.29) | 22.55 (45.41)

12. Secondary Outcome: Change in Status of the Subject (Off) After Wake-up From Baseline to the End of Double-blind Maintenance Period
Description: A subject has been considered "off" when he/she began to lose the optimum effects of anti-Parkinson's medication.
  The percentage of days from Baseline to the end of the double-blind Maintenance Period in which the subject woke in the "off" state is presented below.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
percentage of days | -10.34 (47.81) | -21.14 (48.49)

13. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS Part III Motor Examination) During "on" Periods From Baseline to the End of Double-blind Maintenance Period
Description: The UPDRS Part III (motor subscale) assessment consists of 27 questions, measured on a 5-Point scale (0 to 4). The sum score is calculated as sum of these 27 individual questions. This score ranges from 0 to 108, higher scores denote greater disability.
  A subject has been considered "on" when he/she felt the effects of L-dopa. The subject recorded the exact time of L-dopa intake and his/her status at the time of the L-dopa dose. In instances when the subject was 'off' when taking his/her L-dopa, he/she recorded the exact time their status changed to 'on'.
Time Frame: From Baseline (Week 0) to end of Maintenance Period (up to Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Full Analysis Set (Placebo Treated Subjects) | Full Analysis Set (Rotigotine Treated Subjects)
Number analyzed (Participants) | 168 | 170
units on a scale | -3.6 (9.8) | -10.4 (10.4)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAE) were collected during the study, which began in August 2012 and concluded in October 2014.
Description: TEAEs are comprised of the Safety Population (SS), which consists of all randomized subjects who received at least 1 dose of study medication.
Groups:
- Placebo: Placebo, daily doses, placebo Group
  Subjects randomized to placebo will receive matching placebo patches.
- Rotigotine: Rotigotine, daily doses, treatment Group
  Subjects will receive rotigotine or placebo patches in escalating weekly doses (starting with daily doses of rotigotine 4 mg/ 24 h or matching placebo) until an optimal dose or maximal dose of rotigotine 16 mg/ 24 h or matching placebo is achieved. A combination of patches (rotigotine or matching placebo) will be applied for subjects who require a dose > 8 mg/ 24 h. Each dose level is maintained for 1 week.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 6/172 | 6/174
Other Adverse Events (participants affected / at risk) | 24/172 | 54/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | Rotigotine (N=174)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=172) | Rotigotine (N=174)
Nausea (Gastrointestinal disorders) | 2 (2) | 16 (23)
Dyskinesia (Nervous system disorders) | 7 (7) | 11 (13)
Dizziness (Nervous system disorders) | 7 (8) | 19 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (11) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.